CLINICAL TRIAL: NCT04537221
Title: Nordic Cystectomy Study III - Prospective Validation of Transfusions as a Poor Prognostic Factor After Radical Cystectomy for Bladder Cancer
Brief Title: Nordic Cystectomy Study III - Transfusion
Acronym: NorCys-Transf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Nordic Urothelial Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: T199/2020
Record Dates: First submitted 2020-08-19; First posted 2020-09-03 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Bladder Cancer; Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No transfusions: Patients receiving no perioperative blood transfusions (PBT)
  Interventions: Biological: Blood transfusion
- Transfusions: Patients receiving perioperative blood transfusions (PBT)
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — Transfusion of red blood cells peri-operatively

SUMMARY:
Around 7200 cases of Muscle Invasive Bladder Cancer are diagnosed annually in the Nordic countries combined. Muscle Invasive Bladder Cancer is an aggressive disease and it is linked with high mortality rates. The golden standard of treatment is radical cystectomy (RC) (the surgical removal of the bladder) and radical removal of lymph nodes in the pelvis. In addition to surgical treatment, and especially in cases where the tumour invades tissues surrounding the bladder or lymph nodes, chemotherapy is recommended. Chemotherapy can be administered before or after surgery, in a neoadjuvant (NAC) or adjuvant setting (AC). Although most patients recover well from surgery, there are significant risks regarding radical cystectomy. The greatest challenges in planning the treatment are making individual risk assessments and prognosis for the treated patients. Neoadjuvant chemotherapy is also insufficiently used and it is hard to predict how the tumour responds to chemotherapy.

The purpose of this study is to collect prospective clinical data on radical cystectomy -patients in co-operation with other Nordic countries: Sweden, Denmark, Iceland and Norway. The collected data is used to validate existing prediction tools and discover novel tools for prediction of morbidity related to RC and prediction of oncological outcome after RC. The study is divided into three sub-studies. Transfusions during RC and the time of hospitalization after the surgery are associated poorer oncological outcome when compared to those patients who do not need transfusions. The third study focuses on the oncological outcomes in patients receiving blood transfusions. As there are some conflicting reports and the finding is not properly validated, we aim to validate the effect of transfusions on survival after RC.

The number of transfusions during RC and the time between surgery and discharge from hospital will be recorded. Patient cohort will be divided into patients receiving transfusions and not receiving transfusion. The primary end point is patients receiving transfusion and its effect on cancer specific mortality at 24 months. For patients receiving NAC, additional secondary end-point is complete response (pT0N0) rate at RC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed urinary BC planned to be treated with RC with or without neoadjuvant chemotherapy.
* Histologically confirmed urinary BC planned to be treated with palliative cystectomy
* Signed informed consent
* Patient age >18 years

Exclusion Criteria:

* RC for other reasons than BC
* Other forms of surgical treatment of BC than RC (e.g. bladder resection).
* Patient unwillingness to participate in the study for any reason (i.e. lack of signed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with muscle-invasive bladder cancer undergoing radical cystectomy -surgery
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood transfusion (PBT) effect on cancer specific mortality | 24 months
  Comparison of cancer-specific-mortality between patients receiving one or more PBT perioperatively vs. patients receiving none

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- University Hospital of Turku, Hospital Distric of Southwest Finland, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No